CLINICAL TRIAL: NCT04830280
Title: The Effect of Ultrasound-guided Posterior Quadratus Lumborum Block on Atelectasis in Pediatric Patients
Brief Title: Effect Posterior QLB on Atelectasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Çağdaş Baytar, medical doctor, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/03-11
Record Dates: First submitted 2021-03-29; First posted 2021-04-05 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Atelectasis; Block; Pediatrics; Quadratus Lumborum Block
Keywords: postoperative atelectasis; ultrasound; lung ultrasound score; posterior QLB
MeSH Terms: conditions — Pulmonary Atelectasis; Bites and Stings

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior quadratus lumborum block (Active Comparator)
  Interventions: Procedure: posterior quadratus lumborum block
- control group (Sham Comparator)
  Interventions: Procedure: posterior quadratus lumborum block

INTERVENTIONS:
Procedure: posterior quadratus lumborum block — administration local anesthetic solution between the middle layer of the thoracolumbar fascia and QL muscle at the posterior edge of the quadratus lumborum muscle

SUMMARY:
We aimed to investigate the effect of posterior quadratus lumborum block on postoperative atelectasis in inguinal hernia surgery in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* under 2 years old,
* ASA I-II risk group
* Patients who underwent an inguinal hernia operation under general anesthesia, posterior quadratus lumborum block for postoperative analgesia or pain treatment with conventional method
* Patients whose informed consent was read and approval was obtained from him and his guardian

Exclusion Criteria:

* who do not want to participate in the study,
* ASA III-IV-V patients

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
lung ultrasound score | up to 1 hour after surgery
  atelectasis

SECONDARY OUTCOMES:
pain scores | up to 6 hour after surgery
  Flacc scores

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No